CLINICAL TRIAL: NCT00719719
Title: Studies in the Pathogenesis of Anaphylaxis
Brief Title: Cause of Unexplained Anaphylaxis
Status: Active, not recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080184; 08-I-0184
Record Dates: First submitted 2008-07-19; First posted 2008-07-22 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-11-19

CONDITIONS: Idiopathic Anaphylaxis; Drug Anaphylaxis; Venom Anaphylaxis; Food Anaphylaxis
Keywords: Antigen Specific; Mast Cell; Tryptase; Bone Marrow; Hives; Natural History; Anaphylaxis
MeSH Terms: conditions — Urticaria; Anaphylaxis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Drug Anaphylaxis: Drug Anaphylaxis
- Food Anaphylaxis: Food Anaphylaxis
- Idiopathic Anaphylaxis: Idiopathic Anaphylaxis
- Venom Anaphylaxis: Venom Anaphylaxis

SUMMARY:
This study will explore the possible cause of unexplained, or idiopathic, anaphylaxis. Anaphylaxis is a rapid, life-threatening, severe reaction that occurs suddenly after contact with an allergy-causing substance, usually a particular food, drug or stinging insect. The allergen triggers mast cells to release several substances, including histamine. Histamine is responsible for many of the symptoms that may occur, such as flushing, hives, swelling of the palms and soles or tongue and vocal cords, nasal congestion, itching and tearing of the eyes, shortness of breath and wheezing, stomach pain, vomiting, low blood pressure, loss of consciousness, shock, and, rarely, death. Severe episodes of anaphylaxis are treated with epinephrine (adrenaline), followed by oral antihistamines and steroids. In more than half of cases of anaphylaxis, a clear cause is not identified. These cases are called idiopathic anaphylaxis. There is no cure or long-term preventive therapy for patients with recurrent episodes of idiopathic anaphylaxis.

People between 13 and 70 years of age who have idiopathic anaphylaxis, or have anaphylaxis that is caused by specific allergens such as food, venom, or drugs and medications may be eligible for this study.

Participants are evaluated at the NIH Clinical Center with the following tests and procedures:

* Medical history, physical examination and blood tests.
* Bone marrow biopsy. For this test, the skin over the hipbone and the outer surface of the hipbone itself are numbed with local anesthesia. Then, a needle is inserted into the hipbone and a small amount of bone marrow is drawn into a syringe. The needle also cuts a small core of bone marrow, which is removed for analysis.
* Other tests that may be needed for evaluation of the patient s condition.

DETAILED DESCRIPTION:
Anaphylaxis is a severe life-threatening systemic hypersensitivity reaction caused by release of mediators from mast cells and basophils, characterized by cutaneous, respiratory, cardiovascular, or gastrointestinal signs and symptoms. The most common specific causes of anaphylaxis are venom, drug, and food allergies (i.e. patients with specific anaphylaxis, SA), When a causative factor is not identified in patients are said to have idiopathic anaphylaxis (IA). Evidence of an underlying clonal mast cell disease has been found in about I in 15 patients with IA in our studies and in about 1 in 12 patientswith venom induced anaphylaxis in a European study. (1) The number of patients with anaphylaxis to foods or drugs who have a clonal mast cell disease is not known and the number or patients with venom induced anaphylaxis in the US with clonal mast cell disease has not been determined. Thus, a more complete understanding of the prevalence of clonal mast cell disease in those experiencing anaphylaxis and a better understanding of the associated laboratory abnormalities and disrupted molecular signaling pathways will have a substantial impact of the clinical management of patients who present with anaphylaxis.

This protocol thus focuses on determining the prevalence of clonal mast cell disorders in patients with the anaphylaxis, whether unexplained (IA) or associated with exposure to an antigen (SA), and attendant changes in the mast cell compartment. Subjects 13 - 75 years old will be evaluated to correlate both clinical and laboratory features of anaphylaxis and to identify genetic and molecular pathways that may predispose to these events. Subjects may undergo bone marrow examination in addition to supporting laboratory studies when indicated. We plan to enroll up to 200 subjects.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subjects must be at least 13 years of age and no older than 75 years of age.
* Subjects with IA must have a diagnosis of anaphylaxis occurring in the absence of an identifiable provoking agent or stimulus by a referral provider. Patient may carry both the diagnosis of 1A and the diagnosis of SA.
* Subjects with SA must have a history of a severe reaction to a venom, food or, drug confirmed when possible by relevant skin testing, challenge testing, RAST, immunoCAP, or ELISA. within the past 36 months.
* Subject must have had a doctor s office or ER visit, or a hospitalization for evaluation for anaphylaxis and have a history of involvement of the skin and/or mucosal tissue (e.g., flushing, itching, hives, angioedema, tongue swelling), and at least one of the following:

  * Respiratory compromise (e.g., dyspnea, hoarseness-laryngeal edema, wheeze-bronchospasm, stridor, reduced peak expiratory flow, hypoxemia).
  * Gastrointestinal symptoms of vomiting and/or diarrhea
  * Reduced blood pressure and/or associated symptoms of end-organ dysfunction (as evidenced hypotonia, hypoxia, collapse, syncope or incontinence).
* Letter of referral from prospective study participant's referring physician, or similar primary provider - with copies of available medical evaluation and laboratory studies
* Able and willing to consider a bone marrow biopsy and aspirate

EXCLUSION CRITERIA:

* Presence of conditions which in the judgment of the investigator or the referring physician may put the subject at undue risk for travel (including frequent episodes of IA not preventable by pre-medication, acute infection, severe thrombocytopenia [minimum platelet count of 30,000], or significant cardiovascular disease)
* Any condition that - in the view of the principal investigator would make the subject unsuitable for enrollment in this study
* Inability to provide informed consent
* Pregnancy

Ages: 13 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary Clinical
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2008-11-05 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to determine if patients with anaphylaxis (IA or SA) have clinical & laboratory features that correlate with genetic or molecular abnormalities in their mast cell population including the presence o... | 12/31/2028
  The primary objective of this study is to determine if patients with anaphylaxis (IA or SA) have clinical & laboratory features that correlate with genetic or molecular abnormalities in their mast cell population including the presence of clonal mast cell disease.

SECONDARY OUTCOMES:
Explore abnormalities in signaling Evaluate growth and degranulation of mast cells grown in vitro. Identify patients with the D816V mutation | 12/31/2028
  Explore abnormalities in signaling Evaluate growth and degranulation of mast cells grown in vitro. Identify patients with the D816V mutation

CONTACTS AND LOCATIONS:
Overall Officials: Melody C Carter, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
The initial hypothesis for this protocol has already been explored and published. The ongoing hypothesis generated with the expansion of the protocol is ongoing and once data collection is at a level for analysis, we will include in the IPD.

REFERENCES:
- [Background] Sampson HA, Munoz-Furlong A, Campbell RL, Adkinson NF Jr, Bock SA, Branum A, Brown SG, Camargo CA Jr, Cydulka R, Galli SJ, Gidudu J, Gruchalla RS, Harlor AD Jr, Hepner DL, Lewis LM, Lieberman PL, Metcalfe DD, O'Connor R, Muraro A, Rudman A, Schmitt C, Scherrer D, Simons FE, Thomas S, Wood JP, Decker WW. Second symposium on the definition and management of anaphylaxis: summary report--second National Institute of Allergy and Infectious Disease/Food Allergy and Anaphylaxis Network symposium. Ann Emerg Med. 2006 Apr;47(4):373-80. doi: 10.1016/j.annemergmed.2006.01.018. PMID 16546624
- [Background] Webb LM, Lieberman P. Anaphylaxis: a review of 601 cases. Ann Allergy Asthma Immunol. 2006 Jul;97(1):39-43. doi: 10.1016/S1081-1206(10)61367-1. PMID 16892779
- [Background] Patterson R, Hogan MB, Yarnold PR, Harris KE. Idiopathic anaphylaxis. An attempt to estimate the incidence in the United States. Arch Intern Med. 1995 Apr 24;155(8):869-71. doi: 10.1001/archinte.155.8.869. PMID 7717796
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2008-I-0184.html